CLINICAL TRIAL: NCT01257412
Title: A 24-week National Multicenter, Randomized, Double-Blind, Placebo-Controlled, Parallel-Group, Phase III Trial in India to Evaluate the Efficacy and Safety of Dapagliflozin as Monotherapy in Subjects With Type 2 Diabetes Who Have Inadequate Glycaemic Control With Diet and Exercise Alone.
Brief Title: Evaluation of Efficacy and Safety of Dapagliflozin as Monotherapy in Subjects With Type 2 Diabetes Who Have Inadequate Glycaemic Control With Diet and Exercise Alone
Status: Suspended | Phase: Phase 3 | Type: Interventional
Why Stopped: FSI delayed until 15 January 2013
Sponsor: AstraZeneca (Industry)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D1693C00002
Record Dates: First submitted 2010-12-08; First posted 2010-12-09 (Estimated); Last update posted 2012-03-01 (Estimated); Status verified 2012-02

CONDITIONS: Type 2 Diabetes
Keywords: Phase III; Type 2 Diabetes Mellitus; inadequate glycaemic control
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — dapagliflozin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental)
  Interventions: Drug: Dapagliflozin
- 2 (Experimental)
  Interventions: Drug: Dapagliflozin
- 3 (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Dapagliflozin — 5mg Oral dose od
  Arms: 1
Drug: Dapagliflozin — 10 mg Oral dose od
  Arms: 2
Drug: placebo — 5/10 mg Oral dose od
  Arms: 3

SUMMARY:
This study intends to compare the efficacy and safety of dapagliflozin versus placebo in treatment-naïve subjects with type 2 diabetes who have inadequate glycaemic control with diet and exercise alone.

ELIGIBILITY:
Inclusion Criteria:

* Provision of informed consent before participating in the study
* Diagnosed with type 2 diabetes (high blood sugar); HbA1c ≥ 7.2% and ≤10.0%
* Subjects should be drug naïve
* Women of childbearing potential who comply to use an adequate method of contraception to avoid pregnancy throughout the study & who have a negative serum or urine pregnancy test

Exclusion Criteria:

* Subjects received Insulin therapy within one year of enrollment
* Subjects who have severe uncontrolled hypertension
* Subjects who have history of unstable or rapidly progressing renal disease
* Subjects who have severe liver disease
* Subjects who receiving treatment for Human immunodeficiency virus (HIV)

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 375 (Estimated)
Dates: Start 2012-01; Primary Completion 2013-06 (Estimated); Study Completion 2013-06 (Estimated)

PRIMARY OUTCOMES:
change in glycosylated haemoglobin A1c (HbA1c). | From baseline to week 24

SECONDARY OUTCOMES:
mean change in fasting plasma glucose (FPG) | From baseline to week 24
mean change in 2- hour postprandial glucose by Mixed Meal Test | From baseline to week 24
mean change from baseline in fasting plasma glucose (FPG) | From baseline to week 1

CONTACTS AND LOCATIONS:
Overall Officials: Prof. A. Ramachandran, MD, PhD, Principal Investigator — Dr. A. Ramachandran's Diabetes Hospital
Locations (15):
- India (15):
  - Research Site, Hyderabad, Andhra Pradesh
  - Research Site, Vijaywada, Andhra Pradesh
  - Research Site, Ahmedabad, Gujarat
  - Research Site, Bangalore, Karnataka
  - Research Site, Mysore, Karnataka
  - Research Site, Trivandrum, Kerala
  - Research Site, Indore, Madhya Pradesh
  - Research Site, Mumbai, Maharashtra
  - Research Site, Nagpur, Maharashtra
  - Research Site, Pune, Maharashtra
  - Research Site, Jaipur, Rajasthan
  - Research Site, Chennai, Tamil Nadu
  - Research Site, Coimbatore, Tamil Nadu
  - Research Site, Madurai, Tamil Nadu
  - Research Site, Ghaziabad, Uttar Pradesh